CLINICAL TRIAL: NCT06988839
Title: Patient-Centered And Clinical Outcomes Of Microneedling With Coronally Advanced Flap For Management of RT1 Gingival Recession In Thin Gingival Phenotype : A Randomized Controlled Clinical Trial
Brief Title: Effect Of Microneedling With Coronally Advanced Flap For Management of RT1 Gingival Recession In Thin Gingival Phenotype
Acronym: RT1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KASHISH PERIO 25/33
Record Dates: First submitted 2025-05-13; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Gingival Recession
Keywords: gingival recession; percutaneous collagen induction; root coverage; connective tissue graft; microneedle
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedling with coronally advanced flap (Experimental): In this group, microneedling will be performed using a 30 gauge lancet needles, inserted until hard tissue is felt. It will be performed in 4 sessions at 10 day intervals, followed by coronally advanced flap procedure, 2 months post microneedling.
  Interventions: Procedure: Microneedling followed by coronally advanced flap
- Coronally advanced flap with connective tissue graft (Active Comparator): Coronally advanced flap operation will be performed with connective tissue graft harvested from palate after phase 1 therapy.
  Interventions: Procedure: Coronally advanced flap with connective tissue graft

INTERVENTIONS:
Procedure: Microneedling followed by coronally advanced flap — Microneedling will be performed using a 30 gauge lancet needles, inserted until hard tissue is felt. It will be performed in 4 sessions at 10 day intervals, followed by coronally advanced flap procedure, 2 months post microneedling.
  Arms: Microneedling with coronally advanced flap
Procedure: Coronally advanced flap with connective tissue graft — Coronally advanced flap operation will be performed with connective tissue graft harvested from palate after phase 1 therapy.
  Arms: Coronally advanced flap with connective tissue graft

SUMMARY:
The goal of this clinical trial is to explore the effect of microneedling to increase the gingival tissue thickness which could improve the outcome of root coverage in coronally advanced flap procedure in thin gingival phenotype. The main question it aims to answer is that :

Does the use of microneedling procedure followed by coronally advanced flap has similar outcomes of root coverage in recession type 1 (RT1) gingival recession i.e. buccal gingival recessions without interdental clinical attachment loss in thin gingival phenotype as compared to coronally advanced flaps with connective tissue graft.

Systemically healthy patients having isolated upper RT1 gingival recession will be assigned into two groups. Microneedling will be performed in one group (4 sessions each at a 10 days interval) followed by coronally advanced flap operation (at an interval of 2 months) and coronally advanced flap with connective tissue graft will be performed in the other group. Follow-up will be done at 1 month, 3 months and 6 months for evaluation of primary and secondary outcomes.

DETAILED DESCRIPTION:
The gingival phenotype affects the choice of mucogingival surgical technique for coverage of the root surface in gingival recession. It has been reported that a flap thickness of > 0.8 mm results in a covered root surface of 100%, whereas a flap thickness of < 0.8 mm results in partial root coverage in coronally advanced flap procedure for Miller class I or II root coverage. Thus connective tissue graft (CTG) use is advocated in thin phenotype cases, for improved clinical and esthetic outcomes. Connective tissue graft increases the predictability of coronally advanced flap. Treatment by addition of connective tissue graft has some drawbacks like creation of a second surgical site, postoperative discomfort and long chair side time, leading the researchers to explore techniques less invasive in nature.

Microneedling (MN), also known as "percutaneous collagen induction therapy." It creates microinjuries that result in minimal superficial bleedings and create a wound-healing cascade from which various growth factors, such as platelet-derived growth factors, transforming growth factors, connective tissue growth factor and fibroblast growth factors, are released. In microneedling, the tissue responds as if experiencing minor trauma and the body's own collagen production is induced to preserve skin integrity. Microneedling as opposed to connective tissue grafts is a non-surgical approach to increase gingival thickness, that results in significant changes in the gingival thickness and keratinized tissue width of individuals with thin gingival phenotype. It is associated with higher patient acceptance, lesser surgical site co-morbidities and is a minimally invasive yet an effective approach to augment the gingiva. The histological analysis performed one year post microneedling sessions, showed increased collagen and elastic fiber accumulation in the reticular dermis, a thickened epidermis and a normal stratum corneum, showing its greater effect on gingival thickness.

The present study aims to increase the gingival thickness by microneedling procedures to enhance root coverage by coronally advanced flap procedures in thin gingival phenotype. This technique is proposed to improve thin gingival phenotype by minimally invasive and non-surgical means.

ELIGIBILITY:
Inclusion Criteria:

* Presence of isolated RT1 buccal maxillary gingival recessions in esthetic zone with thin gingival phenotype (Gingival thickness≤1mm) associated with esthetic complaints and/or dental sensitivity and otherwise systemically healthy.
* Gingival Recession ≥2mm , Keratinized tissue width≥2mm and clinically identifiable cementoenamel junction
* Age 20years-50 years
* Patient demonstrating compliance for maintaining good oral hygiene after Phase 1 therapy Plaque index (PI) <1, Gingival Index (GI) <1
* Providing a written and verbal informed consent.

Exclusion Criteria:

* Patient with systemic disease that can influence the outcome of therapy.
* Pregnant females or on oral contraceptive pills or hormone replacement therapy.
* Smokers and patients undergoing orthodontic therapy
* Physically and mentally impaired patients.
* Non vital, malpositioned tooth
* Presence of cervical abrasions or restorations in the area
* Previous history of periodontal surgery on the involved sites.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recession depth (RD) | Baseline,1,3,6 months
  It will be recorded in mm with a periodontal probe from the CEJ to the crest of the gingival margin at the mid-labial region
Recession width (RW) | Baseline, 1 , 3 and 6 months
  It will be recorded in mm with a periodontal probe from the mesial to distal gingival margin at the level of cementoenamel junction.
Root coverage percentage (RC%) | Baseline ,1,3 and 6 months
  It will be calculated according to formula Root coverage percentage= RD (preop -postop) *100 /RD preoperative
Root Esthetic Score (RES) | Baseline, 6 months
  The RES system evaluates 5 variables 6 months following surgery: gingival margin, marginal tissue contour (MTC), soft tissue texture (STT), Mucogingival junction alignment, and gingival color (GC). 0, 3, or 6 points will be used for the position of the gingival margin, whereas a score of 0 or 1 point will be used for each of the other variables
Patient-centered outcomes | Baseline,1,3 and 6 months
  Each patient will be questioned about his/her satisfaction with regard to following criteria: root coverage attained, dentinal hypersensitivity, shape and contour of gums, surgical procedure, and post-surgical phase and it will be assessed using a three-point rating scale.

SECONDARY OUTCOMES:
Clinical Attachment level (CAL) | Baseline, 1 , 3 ,6 months
  Clinical attachment level will be measured as the distance between the CEJ and the base of pocket. Measurements will be made at 6 sites of each tooth using periodontal probe.
Probing pocket depth | Baseline,1 ,3 and 6 months
  Probing pocket depth will be measured as the distance from gingival margin to the base of pocket. Measurements will be noted at 6 sites of a tooth.
Plaque index | Baseline, 1 ,3 and 6 months
  Plaque index will be measured on buccal and lingual surface with Periodontal probe.
Gingival index | Baseline,1,3 and 6 months
  Gingival index will be used to assess severity of gingival inflammation with the help of periodontal probe at 4 sites.
Gingival thickness | Baeline, 1 ,3 and 6 months
  A No:15 endodontic spreader with silicon disc as stopper will be inserted perpendicularly at 1.5mm apical to gingival margin, till the hard tissue will be felt. The depth of penetration will be noted using digital calliper measuring the distance between the tip of the spreader and silicon disc.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No